CLINICAL TRIAL: NCT00290914
Title: Safety and Efficacy Study of Vilazodone and Discovering Genetic Markers Associated With Response in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacology Research Institute (Other)
Purpose: Treatment
Other Study IDs: PRI #608
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vilazodone Hydrochloride

INTERVENTIONS:
Drug: Vilazodone

SUMMARY:
The purpose is to evaluate the safety and usefulness of the investigational drug, vilazodone in depression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18-65 years of age, inclusive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult